CLINICAL TRIAL: NCT01399346
Title: A Single-center, Randomized, Controlled, 2-period Cross-over, Open-labelled Trial to Evaluate the Impact of Different Application Volumes on Pharmacokinetic and Pharmacodynamic Properties of Insulin Aspart in Subjects With Type 1 Diabetes
Brief Title: Investigation of the Impact of Different Application Volumes of Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Pieber Thomas, MD, MD, Prof. of Medicine, Medical University of Graz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SPRINK-01
Record Dates: First submitted 2011-05-23; First posted 2011-07-21 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Type 1 Diabetes
Keywords: Insulin aspart; Type 1 diabetes; Glucose clamp; Pharmacodynamics; Pharmacokinetics; Rapid Acting Insulin Analog
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 bolus of insulin aspart 18 IU (Experimental): Subcutaneous administration of insulin aspart as one bolus of 18 IU at one injection site.
  Interventions: Drug: Insulin aspart
- 9 bolus of insulin aspart a 2 IU (Experimental): Subcutaneous administration of insulin aspart as 9 separately and simultaneously applied bolus of 2 IU at 9 separate injection sites
  Interventions: Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin aspart — Application of 18 IU insulin aspart as one bolus at one injection site
  Arms: 1 bolus of insulin aspart 18 IU
Drug: Insulin aspart — Application of 18 IU insulin aspart as 9 bolus of 2 IU each at nine injection sites
  Arms: 9 bolus of insulin aspart a 2 IU

SUMMARY:
Rationale: For the development of a closed loop system, faster insulin absorption after bolus administration could help to reduce the system's delay and thus increase patient safety. It has been shown that regular insulin absorption is faster when injecting insulin with a sprinkler needle (containing holes in the walls and being sealed at the tip). The current study will evaluate the impact of different application volumes on pharmacokinetic and pharmacodynamic properties of rapid acting insulin analogue (insulin aspart).

Objective: To compare the pharmacokinetic response (based on the time to maximum observed serum insulin concentration) and pharmacodynamic properties of rapid acting insulin aspart after subcutaneous injection of a defined dose (volume) at 1 versus 9 injection sites in patients with type 1 diabetes.

Study design: Monocentric, randomised, controlled, two-arm cross-over intervention study.

Population: Twelve type 1 diabetic subjects

Intervention: The investigational treatment is the subcutaneous administration of insulin aspart either as one bolus of 18 IU at one injection site or as 9 separately and simultaneously applied bolus of 2 IU each at 9 separate injection sites. Serum and plasma samples to assess pharmacodynamic and pharmacokinetic properties will be taken during an 8-hour clamp experiment. Patients will undergo both investigational treatments in a randomized order; between the two clamp visits there will be a wash-out period of 5-21 days.

Main study endpoint: Time to maximum observed serum insulin aspart concentration.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged 18-60 years (both inclusive)
* Type 1 diabetes treated with multiple daily insulin injection or continuous subcutaneous insulin infusion for 12 months
* Fasting C-peptide < 0.3nmol/L
* Body mass index 20.0-28.0 kg/m² (both inclusive)
* HbA1c < 10%

Exclusion Criteria:

* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods
* Skin pathology or condition prohibiting needle insertion/insulin administration as judged by the investigator
* History of bleeding disorder
* Current participation in another clinical study
* Significant acute or chronic illness that might interfere with subject safety or integrity of results as judged by the investigator
* Smoker (defined as >5 cigarettes/d)
* Lipodystrophy
* Current treatment with systemic (oral or i.v.) corticosteroids, monoamine oxidase (MAO) inhibitors, non-selective beta-blockers, growth hormone, herbal products or non-routine vitamins. Furthermore, thyroid hormones are not allowed unless the use of these has been stable during the past 3 months.
* Significant history of alcoholism or drug abuse or a positive result in urine drug/alcohol screen.

Study Day Exclusion Criteria:

* Strenuous exercise within the last 24 hours prior to dosing.
* Non-fasting (i.e. consumption of food or beverages, other than water, later than 22:00 hours the evening before the visit) except if slight intake of rapidly absorbable carbohydrates has been necessary in order to prevent hypoglycaemia.
* Injection of long-acting insulin (e.g. insulin glargine or insulin detemir) later than 12:00 hours (noon), 2 days before the dosing visit.
* Injection of NPH insulin or other intermediate-acting insulin products later than 12:00 hours (noon) on the day before the dosing visit.
* Injection of any short acting insulin (aspart, lispro, glulisine) or more than 6 IU of human insulin between 22:00 hours and 03:00 hours the night before the dosing visit.
* Injection of any insulin later than 03:00 hours the night before the dosing visit.
* Infusion of any insulin later than 03:00 hours the night before the dosing visit for subjects using continuous subcutaneous insulin infusion (CSII).
* Positive result of alcohol breath test.
* Any medical condition that, in the opinion of the Investigator, could interfere with insulin pharmacokinetics and/or glucose metabolism.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
tmax(ins), time to maximum observed serum insulin aspart concentration | 8 hours

SECONDARY OUTCOMES:
t10%max(ins), time to reach 10% of maximum observed serum insulin aspart concentration | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- See also: Medical University of Graz — http://www.medunigraz.at